CLINICAL TRIAL: NCT06614270
Title: Clinical Study of Core Blood-derived Anti-CD19 IL-10/IL15 CAR-NK in the Treatment of Refractory/Relapsed Autoimmune Diseases
Brief Title: Anti-CD19 IL-10/IL15 CAR-NK Cells in Refractory/Relapsed Autoimmune Diseases
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2024-1208
Record Dates: First submitted 2024-09-24; First posted 2024-09-26 (Actual); Last update posted 2025-12-29 (Actual); Status verified 2025-09

CONDITIONS: Systemic Sclerosis (SSc); ANCA Associated Vasculitis (AAV); Idiopathic Inflammatory Myopathy (IIM); Sjogren's Syndrome; Antiphospholipid Syndrome; Systemic Lupus Erythematosus
MeSH Terms: conditions — Scleroderma, Systemic; Anti-Neutrophil Cytoplasmic Antibody-Associated Vasculitis; Myositis; Antiphospholipid Syndrome; Lupus Erythematosus, Systemic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Participant Group (Experimental): Anti-CD19 IL-10/IL15 CAR-NK
  Interventions: Drug: Anti-CD19 IL-10/IL15 CAR-NK

INTERVENTIONS:
Drug: Anti-CD19 IL-10/IL15 CAR-NK — Patients will receive Fludarabine and Cyclophosphamide for conditioning. Multiple doses of Anti-CD19 IL-10/IL15 CAR-NK cells will be infused on Day 0, 3, and 6.

SUMMARY:
This study is a single-center, open-label, single-arm, dose-escalation trial. The aim of this study is to investigate the safety and efficacy of Anti-CD19 IL-10/IL15 CAR-NK cells in patients with refractory/relapsed autoimmune diseases, including systemic lupus erythematosus, systemic sclerosis, idiopathic inflammatory myositis, ANCA associated vasculitis, sjogren syndrome, and antiphospholipid syndrome.

ELIGIBILITY:
Common inlcusion Criteria:

1. Age 18-65 years old, male or female;
2. Routine blood count: hemoglobin ≥60g/L, white blood cell count ≥ 2.5×109/L, neutrophil count ≥1.0×109/L (no colony-stimulating factor treatment within 2 weeks before examination);
3. Liver function: ALT ≤3×ULN, AST≤3×ULN, TBIL≤1.5×ULN;
4. Coagulation function: international normalized ratio (INR) < 1.5×ULN, prothrombin time (PT) <1.5×ULN;
5. Cardiac function: good hemodynamic stability;
6. Female subjects of childbearing age must have a negative pregnancy test and agree to use effective contraception during the trial;
7. Voluntarily participate in this study and sign the informed consent form, agreeing to participate in the follow-up as required.

SLE Enrollment Criteria:

1. patients meet the classification criteria of SLE;
2. Refractory or relapsed cases classified as non-response to standard therapy or disease recurrence after remission. Standard treatment is defined as therapy with at least three agents, including glucocorticoids at a dose >1 mg/kg/day, together with at least two of the following immunomodulatory drugs administered for more than 6 months: cyclophosphamide, mycophenolate mofetil, azathioprine, methotrexate, leflunomide, tacrolimus, cyclosporine, iguratimod, antimalarials, and biologic agents, including rituximab, belimumab, or telitacicept.

Systemic Sclerosis (SSc) Enrollment Criteria:

1. Patients who meet the SSc classification criteria of the 2013 ACR/EULAR and have a diagnosis of systemic sclerosis;
2. the patient's disease duration ≤ 60 months (defined as the onset of the first non-Raynaud's symptoms);
3. Patient-modified Rodnan skin score (mRSS) ≥10 at the baseline visit; or active interstitial lung disease (ILD): ground-glass opacity on high-resolution computed tomography (HRCT), pulmonary function suggestive of forced vital capacity (FVC) or diffusing capacity for carbon monoxide (DLCO) less than 70% predicted;
4. A or B needs to be met:

A. Refractory or relapsed cases classified as non-response to standard therapy or disease recurrence after remission. Standard treatment is defined as the use of glucocorticoids and cyclophosphamide, as well as any of the following immunomodulatory drugs, for more than 6 months: antimalarials, azathioprine, mycophenolate mofetil, methotrexate, leflunomide, tacrolimus, cyclosporine, and biologics including rituximab, belimumab, tocilizumab, etc.; B. Presence of progressive disease, specifically defined as, within the past 6 months: a) Progression of cutaneous involvement: more than 25% increase in mRSS; or b) progression of lung disease: 10% reduction in FVC, or 5% reduction in FVC with 15% reduction in DLCO.

Idiopathic Inflammatory myopathy enrollment criteria:

1. Diagnosis according to the 2017 EULAR/ACR classification criteria for inflammatory myopathies, including dermatomyositis (DM), polymyositis (PM), antisynthetase antibody syndrome (ASS), and immune-mediated necrotizing myositis (IMNM);
2. patients with muscle involvement with a manual strength test-8 (MMT-8) score less than 142 and at least 2 abnormalities in the following 5 core assessments: Physician Global Assessment (PhGA), Patient Global Assessment (PtGA), Extramuscular Disease Activity Score ≥2 points, Health Assessment Questionnaire (HAQ) total score ≥0.25, muscle enzyme level ≥1.5×ULN); or MMT-8≥142 with active interstitial lung disease (HRCT suggests ground-glass opacities);
3. Positive myositis-specific antibodies;
4. A or B needs to be met:

A. Relapsed or refractory patients: relapsed or reactive after remission. Definition of conventional treatment: use of glucocorticoids (more than 1 mg/kg/d) and cyclophosphamide and any one or more of the following immunomodulatory drugs for more than 6 months: antimalarials, azathioprine, mycophenolate mofetil, methotrexate, leflunomide, tacrolimus, cyclosporine, and biologics including rituximab, belimumab, tetatercept, etc.; B. Patients with progressive disease: rapid progressive interstitial pneumonia in a short period of time.

ANCA-associated vasculitis enrollment criteria:

1. Meets the 2022 ACR/EULAR ANCA-ASSOCIATED VASCULITIS CLASSIFICATION CRITERIA, INCLUDING MICROSCOPIC POLYANGIITIS (MPA), GRANULOMATOSIS WITH POLYANGIITIS (MPA);
2. Positive PR3-ANCA or MPO-ANCA (either previous or current positive);
3. Birmingham Vasculitis Activity Scale (BVAS) score of ≥ 15 points, and at least 1 major item caused by active vasculitis, or at least 3 non-major items, or at least renal involvement hematuria, proteinuria;
4. estimated glomerular filtration rate (eGFR) ≥15 mL/minute/1.73 m2 (MDRD method);
5. Definition of refractory/relapsed: Conventional treatment that remains ineffective for more than 6 months, or disease recurrence after remission. Conventional treatment definition: use of glucocorticoids (more than 1 mg/kg/day) and cyclophosphamide, as well as any one or more of the following immunomodulatory drugs: antimalarials, azathioprine, mycophenolate mofetil, methotrexate, leflunomide, tacrolimus, cyclosporine, and biologics including rituximab, belimumab, tocilizumab, etc.

Sjögren's syndrome enrollment criteria:

1. Meet the 2002 European and American Consensus Group (AECG) standards or the 2016 ACR/EULAR Primary Sjögren's Syndrome (pSS) classification criteria;
2. positive anti-SSA/Ro-60 antibody;
3. Definition of disease activity: EULAR Sjögren's Syndrome Disease Activity Index (ESSDAI) score ≥ 5;
4. Definition of recurrence/refractory: Conventional treatment that remains ineffective for more than 6 months, or disease recurrence after remission. Conventional treatment is defined as the use of glucocorticoids (>1 mg/kg/day) and cyclophosphamide, as well as any one or more of the following immunomodulatory drugs: antimalarials, azathioprine, mycophenolate mofetil, methotrexate, leflunomide, tacrolimus, cyclosporine, and biologics including belimumab, rituximab, and tocilizumab.

Antiphospholipid syndrome enrollment criteria:

1. Primary antiphospholipid syndrome meeting the 2006 Sydney criteria;
2. Medium to high titer phospholipid antibody (aPL) positive: lupus anticoagulant (LA), IgG or IgM anti-β2 glycoprotein 1 antibody (anti-β2-GP1) or anticardiolipin antibody (aCL), at least 2 or more times positive, with an interval of more than 12 weeks;
3. A or B needs to be met:

A. Definition of refractory/relapsed: recurrent thrombosis with standard therapy with warfarin or other vitamin K antagonist coagulation (INR maintained within the range required for treatment), or standard therapeutic dose low molecular weight heparin (LMWH) with glucocorticoids and cyclophosphamide; B. Catastrophic antiphospholipid syndrome requires the following four criteria: (1) involvement of ≥ 3 organs, systems, and/or tissues (vascular embolism requires radiographic evidence, renal involvement requires a >50% increase in creatinine, blood pressure > 180/100 mmHg, and/or urine protein >0.5 g/24 hours); (2) all clinical manifestations appear simultaneously or sequentially within 1 week; (3) Pathological basis for the presence of small vessel occlusion in at least one organ or tissue (evidence of vascular embolism is required for pathological diagnosis, occasionally complicated by vasculitic manifestations); (4) Positive aPL antibody.

Common Exclusion Criteria:

1. Combined with other connective tissue diseases;
2. Involvement of important organs: heart (individuals with more severe heart disease, such as angina, myocardial infarction, heart failure, and arrhythmias), kidney (eGFR < 15 ml/min/1.73m2), liver (ALT>3×ULN, AST>3×ULN, TBIL >1.5×ULN), lung (FVC<50% predicted or hemoglobin-corrected DLCO<40% predicted), hematologic (leukocyte < 2.5×109/L, neutrophil count <1.0×109/L, HGB<60g/L), etc.;
3. Abnormal hepatitis B or hepatitis C test indicating active infection or chronic infection, including positive HBsAg or HBcAb test and positive hepatitis C antibody;
4. Have active tuberculosis or latent tuberculosis;
5. Human immunodeficiency virus (HIV) serology positivity or known history of HIV infection;
6. Presence of any known serious active infection (including bacterial, viral, fungal, etc.), including those requiring hospitalization or intravenous antibiotic therapy within 4 weeks prior to screening and oral antibiotic therapy within 2 weeks prior to screening; Those who have various chronic infections and are currently receiving corresponding treatment, such as pneumocystosis, cytomegalovirus, herpes zoster, atypical mycobacteria, etc.;
7. Patients with primary or secondary immunodeficiency;
8. IgA deficiency (<10 mg/dL) or IgG deficiency (<400 mg/dL);
9. Receiving other investigational drug treatment or participating in any other drug trial within 3 months before screening;
10. History of documented and confirmed malignancy within 5 years prior to screening, with the exception of basal cell carcinoma of the skin or carcinoma in situ of the cervix that has been appropriately treated or resected;
11. Patients who are pregnant, breastfeeding, or planning a recent pregnancy, or who are unwilling to use a reliable contraceptive method of contraception for the duration of the study;
12. Those who have been allergic to human or murine proteins and monoclonal antibodies in the past;
13. Received live vaccine or live attenuated vaccine within 4 weeks prior to randomization;
14. Patients who are not expected to comply with the requirements of the protocol or are not expected to complete the trial as planned (such as those with psychiatric disorders, history of alcoholism, drug or other substance abuse);
15. Other conditions that the investigator considers the patient not suitable to enter the trial.

Systemic Sclerosis Exclusion Criteria:

1. Localized cutaneous SSc;
2. the duration of the disease is greater than 5 years (defined as the onset of the first non-RP symptom);
3. SSc-like syndrome related to environmental factors, such as vinyl chloride, bleomycin, etc.;
4. Any history of scleroderma renal crisis;
5. intermediate- and high-risk pulmonary hypertension;
6. Active antral vasodilation.

Idiopathic Inflammatory myopathy exclusion criteria:

1. drug-induced myopathy;
2. inclusion body myositis;
3. Tumor-associated myositis (myositis occurring within 2 years of diagnosis of tumor).

ANCA-associated vasculitis exclusion criteria:

1. alveolar hemorrhage, requiring invasive lung ventilation, which is expected to last longer than the screening time;
2. Need for dialysis or plasmapheresis during screening;
3. Have undergone a kidney transplant.

Sjögren's syndrome exclusion criteria:

1. Combined with liver cirrhosis;
2. Combined with aplastic anemia (AA), myelodysplastic syndrome (MDS) or other myeloproliferative disorders (MPD);
3. drug-induced thrombocytopenia;
4. Thrombotic thrombocytopenic purpura (TTP)/microthrombotic vascular disease (TMA).

Antiphospholipid syndrome exclusion criteria:

1. Obstetric APS;
2. APS incorporates other CTDs;
3. APS involves the nervous system.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2025-01-06 (Actual); Primary Completion 2026-01-06 (Estimated); Study Completion 2027-01-06 (Estimated)

PRIMARY OUTCOMES:
The proportion of subjects with DLT | Within 28 days after anti-CD19 CAR-NK cells infusion
  DLT definition is dose-limiting toxicity.
The proportion of subjects with adverse events | 12 months
  Incidence and severity of AEs and SAEs, including changes in laboratory values, ECG and vital signs as assessed by CTCAE v5.0.

SECONDARY OUTCOMES:
Changes in SLEDAI-2K scores and the proportions of patients achieving SRI-4 response, DORIS remission, and LLDAS in systemic lupus erythematosus. | 12 months
changes of mRSS score for systemic sclerosis | 48 weeks
definition of improvement by IMACS for IIM | 48 weeks
STAR score for sjogren's syndrome | 48 weeks
BVAS for AAV | 48 weeks
Thrombosis/death for APS | 48 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- the second affiliated hospital Zhejiang University School of Medicine, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: Undecided